CLINICAL TRIAL: NCT01453764
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intravenously Into Patients With Multiple Sclerosis
Brief Title: Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Into Patients With Multiple Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-MS-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-18 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Nervous System Diseases
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adipose SVF IV Infusion (Experimental): IV Infusion of Autologous Adipose Derived Stromal Vascular Fraction Intervention: Intravenous Infusion
  Interventions: Procedure: Harvesting and Implantation of SVF

INTERVENTIONS:
Procedure: Harvesting and Implantation of SVF — The cell therapy in this study is composed of stem cells derived from a patient's own adipose tissue that are harvested by liposuction using tumescent technique and isolated in the laboratory. The Adipose SVF will be delivered via intravenous injection.

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients with Multiple Sclerosis and clinical outcomes?

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of Adipose-Derived Stromal Cells (ASC) implantation performed intrathecally and intravenously. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Duration of disease: >5 years
* Failure to respond or intolerance to the currently available Multiple Sclerosis (MS) immunomodulatory treatments (ie interferons, Copaxone, immunosuppression): the lack of response to these treatments will be determined/defined by either an increase (deterioration) of at least one degree in the Expanded Disability Status Scale (EDSS) score during the last year or the appearance of at least two major relapses of MS during the same period of time (under treatment) or intolerance to these agents.
* Up to date on all age and gender appropriate cancer screening per American Cancer Society .

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. For patients who have tested positive, an expert will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection.
* Cerebrovascular accident within 6 months prior to study entry
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement in disability score compared to baseline | 3 months
Number of patients with adverse events | up to 6 months
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.
Clinical improvement in disability score compared to baseline | 6 months

SECONDARY OUTCOMES:
MS disease activity measured by the number of Gd-enhancing brain MRI lesions | 3 months
Reduced number of relapses or freedom from progression of disease | 3 months
Reduced number of relapses or freedom from progression of disease | 6 months
MS disease activity measured by the number of Gd-enhancing brain MRI lesions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided